CLINICAL TRIAL: NCT03089749
Title: Characterization of Human Autoantibody Titers After Central Nervous System Insult
Acronym: CHAT CNS
Status: Terminated | Type: Observational
Why Stopped: This study has been administratively closed by the IRB as of 5/20/2019. This administrative closure was required because of the study expiration on 4/29/2019 and a continuing review application for re-approval of the study was not submitted.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: CHAT-00081214
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Brain Injuries, Traumatic; Spinal Cord Trauma; Intracranial Neoplasm
MeSH Terms: conditions — Brain Injuries, Traumatic; Spinal Cord Injuries; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control: Participants with no history of Traumatic Brain Injury, Traumatic Spinal Cord Injury or Intracranial Neoplasm. A single draw of 5 mL of blood will be obtained as well as demographic information and a brief medical history to act as comparison data to the other groups.
- Traumatic Brain Injury (TBI): Patients with Acute Severe TBI (post-resuscitation GCS of 8 or less). Participants will have blood draws at the time points identified below:
  * At 24h from the time of CNS insult
  * At 3, 5, 7, 10, 14, 18, 21, 30 days from the time of CNS insult
  * At 3, 6, and 12 months from the time of CNS insult
  * Annually for the next four years Total of up to 16 blood draws.
  In all cases, 5 mL of blood will be obtained from the participant. Demographic data will be collected, including:
  * Age
  * Sex
  * History of prior CNS insult
  * Clinical indicators of severity including baseline, post-resuscitation Glasgow Coma Scale (GCS) scores for brain injury patients
  * Radiographic indicators of severity including volume of intracranial hemorrhage, effacement of basal cisterns, amount of midline shift as well as Marshall and Rotterdam CT head scores for TBI.
  * Outcome data including discharge, 3-, 6-, and 12-month extended Glasgow Outcome Scale (GOS) scores
- Spinal Cord Injury (SCI): Patients with acute spinal cord injury (SCI) (post-resuscitation ASIA score of C, B or A). Participants will have blood draws at the time points identified below:
  * At 24h from the time of CNS insult
  * At 3, 5, 7, 10, 14, 18, 21, 30 days from the time of CNS insult
  * At 3, 6, and 12 months from the time of CNS insult
  * Annually for the next four years Total of up to 16 blood draws.
  In all cases, 5 mL of blood will be obtained. Demographic data will be collected, including:
  * Age
  * Sex
  * History of prior CNS insult
  * Clinical indicators of severity including baseline post-resuscitation American Spinal Injury Association (ASIA) score and ASIA impairment scale (AIS) grade for patients with spinal cord injury (SCI)
  * Radiographic indicators of severity including the degree of cord compression, area of cord signal change and the SFGH MRI scale will be employed.
  * Outcome data including discharge, 3-, 6-, and 12-month ASIA scores for SCI patients
- Intracranial Neoplasm: Patients undergoing resection of intra-axial brain tumors (commonly gliomas such as glioblastoma multiforme, astrocytomas and oligodendrogliomas). All participants will have blood draws at the time points identified below:
  * At 24h from the time of CNS insult
  * At 3, 5, 7, 10, 14, 18, 21, 30 days from the time of CNS insult
  * At 3, 6, and 12 months from the time of CNS insult
  * Annually for the next four years Total of up to 16 blood draws.
  In all cases, 5 mL of blood will be obtained. Demographic data will be collected, including:
  * Age
  * Sex
  * History of prior CNS insult
  * Clinical indicators of severity including baseline, Karnofsky and Modified Rankin performance status scores for oncology patients.
  * Radiographic indicators of severity including the pre- and postoperative tumor volumes that will be quantitated.
  * Outcome data including discharge, 3-, 6-, and 12-month Karnofsky and Modified Rankin scores for oncology patients.

SUMMARY:
The aim of the study is to quantitate Central Nervous System (CNS) autoantibody development in human blood using ELISA after human brain injury, spinal cord injury, and intra-axial brain surgeries.

DETAILED DESCRIPTION:
Study Objectives:

We aim to:

1. Quantitate CNS autoantibody development in human blood using ELISA after human brain injury, spinal cord injury, and intra-axial brain surgeries. We also aim to characterize the temporal course of this response.
2. Characterize how CNS autoantibody levels correlate with specific injury patterns as well as radiographic and clinical measures of injury severity.
3. Determine how intercurrent infection and a history of prior CNS insult affects the temporal course and magnitude of autoantibody production.

ELIGIBILITY:
Inclusion Criteria:

* Have a severe traumatic brain injury
* Have spinal cord injury ASIA grade A, B or C
* Undergoing resection of intra-axial brain tumors

Exclusion Criteria:

* Participant who is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population includes patients admitted to the University of Utah and its covered entities.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-05; Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Quantitate Autoantibodies | 5 years
  Quantitate CNS autoantibody development and temporal course in human blood using ELISA after human brain injury, spinal cord injury, and intra-axial brain surgeries.

SECONDARY OUTCOMES:
Autoantibody Correlation | 5 years
  Characterize how CNS autoantibody levels correlate with specific injury patterns as well as radiographic and clinical measures of injury severity.
Autoantibody Production and History | 5 years
  Determine how intercurrent infection and a history of prior CNS insult affects the temporal course and magnitude of autoantibody production.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory WJ Hawryluk, MD, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robinson AP, Harp CT, Noronha A, Miller SD. The experimental autoimmune encephalomyelitis (EAE) model of MS: utility for understanding disease pathophysiology and treatment. Handb Clin Neurol. 2014;122:173-89. doi: 10.1016/B978-0-444-52001-2.00008-X. PMID 24507518
- [Background] Becker KJ, Kindrick DL, Lester MP, Shea C, Ye ZC. Sensitization to brain antigens after stroke is augmented by lipopolysaccharide. J Cereb Blood Flow Metab. 2005 Dec;25(12):1634-44. doi: 10.1038/sj.jcbfm.9600160. PMID 15931160
- [Background] Becker KJ, Kalil AJ, Tanzi P, Zierath DK, Savos AV, Gee JM, Hadwin J, Carter KT, Shibata D, Cain KC. Autoimmune responses to the brain after stroke are associated with worse outcome. Stroke. 2011 Oct;42(10):2763-9. doi: 10.1161/STROKEAHA.111.619593. Epub 2011 Jul 28. PMID 21799171
- [Background] Giunta B, Obregon D, Velisetty R, Sanberg PR, Borlongan CV, Tan J. The immunology of traumatic brain injury: a prime target for Alzheimer's disease prevention. J Neuroinflammation. 2012 Aug 1;9:185. doi: 10.1186/1742-2094-9-185. PMID 22849382
- [Background] Noble LJ, Wrathall JR. Distribution and time course of protein extravasation in the rat spinal cord after contusive injury. Brain Res. 1989 Mar 13;482(1):57-66. doi: 10.1016/0006-8993(89)90542-8. PMID 2706482
- [Background] Hayes KC, Hull TC, Delaney GA, Potter PJ, Sequeira KA, Campbell K, Popovich PG. Elevated serum titers of proinflammatory cytokines and CNS autoantibodies in patients with chronic spinal cord injury. J Neurotrauma. 2002 Jun;19(6):753-61. doi: 10.1089/08977150260139129. PMID 12165135